CLINICAL TRIAL: NCT03756558
Title: Cross-SealTM IDE Trial: Prospective, Multi-Center, Single Arm Study of the Cross-SealTM Suture-Mediated Vascular Closure Device System
Brief Title: Cross-Seal Closure Device IDE Trial - Study of the Cross-SealTM Suture-Mediated Vascular Closure Device System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIS2018-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-28 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-06

CONDITIONS: Vascular Closure

STUDY DESIGN:
Intervention Model Description: Performance goal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Cross-Seal System (Experimental): The Cross-Seal System will be used in all subjects enrolled in the study
  Interventions: Device: Cross-Seal System

INTERVENTIONS:
Device: Cross-Seal System — Use of the Cross-Seal system to close the femoral arteriotomy

SUMMARY:
This study evaluates the safety and effectiveness of the Cross-Seal vascular closure device in gaining post procedure hemostasis in subjects undergoing interventional procedures requiring an 8 to 18 french size introducer sheath.

DETAILED DESCRIPTION:
The Cross-Seal device is a VCD intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (8-18F ID) interventional devices. The function of Cross-Seal is to percutaneously close the puncture in the artery wall (arteriotomy) through which the catheters were inserted for the procedure.

The study is being conducted to demonstrate the safety and effectiveness of Cross-Seal in achieving hemostasis in femoral arterial access sites in subjects undergoing percutaneous transcatheter interventional procedures using a large-bore procedure sheath.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject is scheduled for elective or planned (i.e., not emergent or urgent) percutaneous transcatheter interventional procedures involving access through the femoral artery using 8-18 French introducer sheaths
3. Subject is able to undergo emergent vascular surgery if a complication related to the vascular closure necessitates such surgery
4. Subject is willing and able to complete follow-up requirements
5. Subject, or authorized representative signs a written Informed Consent form prior participating in the study

Exclusion Criteria:

General Exclusion Criteria

1. Prior intra-aortic balloon pump at access site
2. Subjects with severe inflow disease (iliac artery diameter stenosis > 50%) and/or severe peripheral arterial disease (Rutherford Classification 5 or 6), as confirmed with prior standard of care Computed Tomography Imaging, duplex ultrasound, and/or intra-procedural fluoroscopy
3. Common femoral artery lumen diameter is < 5 mm
4. In opinion of the investigator, significant scarring of the target access site which would preclude use of the device in accordance with the IFU
5. Prior target artery closure with any closure device < 90 days, or closure with manual compression ≤ 30 days prior to index procedure
6. Prior vascular surgery, vascular graft, or stent in region of access site
7. Subjects receiving glycoprotein IIb/IIIa inhibitors before, during, or after the catheterization procedure
8. Subjects with significant anemia
9. Subject with known bleeding disorder including thrombocytopenia (platelet count < 100,000), thrombasthenia, hemophilia or Von Willebrand's disease
10. Subject with renal insufficiency, on dialysis therapy, or with renal transplant
11. Known severe allergy to contrast reagent that cannot be managed with premedication
12. Inability to tolerate aspirin and/or other anticoagulation/antiplatelet treatment
13. Planned anticoagulation therapy post-procedure such that the Activated Clotting Time (ACT) is expected to be elevated above 350 seconds for more than 24 hours after the procedure
14. Connective tissue disease (e.g., Marfan's Syndrome)
15. Thrombolytics (e.g., streptokinase, urokinase), Angiomax (bivalirudin) or other thrombin-specific anticoagulants ≤ 24 hours prior to the procedure
16. Recent (within 8 weeks) cerebrovascular accident or Q-wave myocardial infarction
17. Subjects who are morbidly obese
18. Planned major intervention or surgery, including planned endovascular procedure in the target leg, within 30 days following the interventional procedure
19. Subject unable to ambulate at baseline (i.e., confined to wheelchair or bed)
20. Currently participating in a clinical study of an investigational device or drug that has not completed its primary study endpoint
21. Known allergy to any device component
22. Subject is known or suspected to be pregnant or lactating
23. Evidence of active systemic or local groin infection
24. Subject has other medical, social or psychological problem that in the opinion of the investigator precludes them from participating
25. Subject is mentally incompetent or a prisoner
26. New York Heart Association (NYHA) Class IV heart failure that is uncontrolled and requires treatment in the Intensive Care Unit within 24 hours prior to the index procedure
27. Left Ventricular Ejection Fraction (LVEF) < 20%
28. Unilateral or bilateral lower extremity amputation
29. Known existing nerve damage in the target leg
30. Subjects who have already participated in this study

    Intra-Procedure Exclusion Criteria
31. Access site above the most inferior border of the inferior epigastric artery (IEA) and/or above the inguinal ligament based upon bony landmarks
32. Access site in the profunda femoris or superficial femoral arteries, or the bifurcation of these vessels
33. Ipsilateral femoral venous sheath during the catheterization procedure
34. Common femoral artery calcium, which is visible with prior Computed Tomography Imaging and/or duplex ultrasound
35. Subject in which there is difficulty inserting the introducer sheath or need for greater than 2 ipsilateral arterial punctures at the start of the catheterization procedure
36. Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
37. Evidence of a pre-existing hematoma (> 1.5 cm in diameter), arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the access site
38. Marked tortuosity (at the investigator's discretion) of the femoral or external iliac artery in the target leg based on prior Computed Tomography imaging, fluoroscopy, and/or duplex ultrasound
39. Angiographic evidence of arterial laceration, dissection, or stenosis in the femoral artery that would preclude use of the investigational device
40. Target arteriotomy >18 French sheath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazin Foteh, MD, Principal Investigator — Cardiothoracic and Vascular Surgeons - Austin; Prakash Krishnan, Principal Investigator — Icahan School of Medicine at Mt Sinai
Locations (20):
- United States (20):
  - Vascular Institute of the Rockies, Denver, Colorado
  - River City Clinical Research, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa Hospital, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rutgers, The State University of New Jersey, Piscataway, New Jersey
  - Mt Sinai Medical Center, New York, New York
  - The Trustees of Columbia University in the City of New York, New York, New York
  - University of Rochester, Rochester, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - INTEGRIS Cardiovascular Physicians, Oklahoma City, Oklahoma
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - North Central Heart, Sioux Falls, South Dakota
  - Holston Valley Medical Center, Kingsport, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - St. David's Heart and Vascular dba Austin heart, Austin, Texas
  - Texas Heart Institute and Baylor St. Luke's Medical Center, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krishnan P, Farhan S, Zidar F, Krajcer Z, Metzger C, Kapadia S, Moore E, Nazif T, Garland T, Zhang M, Khera S, Sharafuddin M, Patel VI, Bacharach JM, Coady P, Schermerhorn ML, Shames ML, Rahimi S, Panneton JM, Elkins C, Foteh M. Cross-Seal IDE Trial: Prospective, Multicenter, Single-Arm Study of the Cross-Seal Suture-Mediated Vascular Closure Device System. Circ Cardiovasc Interv. 2024 Jun;17(6):e013842. doi: 10.1161/CIRCINTERVENTIONS.123.013842. Epub 2024 May 6. PMID 38708595

RESULTS

PARTICIPANT FLOW:
Groups:
- Transfemoral Approach: Closure of Common Femoral Artery site of subjects who have undergone interventional catheterization procedure using 8-18FR ID sheaths.
Period: Overall Study
Arm/Group | Transfemoral Approach
Started | 147
Completed | 142
Not Completed | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 132
  More than one race | 3
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Complications
Description: Freedom from major complications of the target limb. Major Complications include: access site vascular injury that requires surgical intervention, access related lower extremity ischemia, access site infection
Time Frame: 30 days post procedure
Population: Pivotal safety cohort included 96 subjects from the full analysis set, comprising all enrolled and treated subjects who experienced at least one component for the safety endpoint or were follow-up to the lower limit of the follow-up window for each time point. Due to missing data from 8 subjects, the analysis was conducted with 88 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Transfemoral Approach: Closure of common femoral artery site of subjects who have undergone interventional catheterization procedures using 8-18Fr ID sheaths
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 88
Participants | 83

2. Primary Outcome: Mean Time To Hemostasis (TTH)
Description: The mean Time To Hemostasis in the Common Femoral Artery (CFA) of the target limb access site with use of the investigational device.
Time Frame: Index Procedure
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects). Number of participants analyzed is 101 as 9 subjects who had an adjunctive intervention and 4 subjects who did not receive the investigational device.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 101
Minutes | 0.4 (1.4)

3. Secondary Outcome: Freedom From Minor Complications
Description: The freedom from minor complications at the target limb access site. Minor Complications include: pseudoaneurysm at the access site, access site hematoma over 10cm, access site wound dehiscence
Time Frame: 30 days post procedure
Population: Pivotal safety cohort included 96 subjects from full analysis set, comprising all enrolled and treated subjects who experienced at least one component for the safety endpoint or were follow-up to the lower limit of the follow-up window for each time point. Due to missing data from 8 subjects, the analysis was conducted with 88 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 88
Participants | 84

4. Secondary Outcome: Number of Participants With Device Related Complications Within 30 Days Post-procedure
Description: Number of subjects with devices related complications as adjudicated by the Clinical Events Committee.
Time Frame: 30 days post procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 88
Participants | 9

5. Secondary Outcome: Incidence of Adverse Events
Description: Incidence of major and minor Adverse Events (AEs)
Time Frame: 60 days post procedure
Population: Pivotal safety cohort included 96 subjects from full analysis set, comprising all enrolled and treated subjects who experienced at least one component for the safety endpoint or were follow-up to the lower limit of the follow-up window for each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 96
Participants | 62

6. Secondary Outcome: Incidence of Technical Success
Description: Incidence of hemostasis with the investigational device without the need for any access-site-related adjunctive surgical or endovascular intervention (target limb only).
Time Frame: Immediately Post-procedure (procedure approximately 8 hours)
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects). Due to missing data from 4 subjects, the analysis was conducted on 110 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Transfemoral Approach: Closure of Common Femoral Artery site of subjects who have undergone interventional catheterization procedures using 8-18Fr ID
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 110
Participants | 102

7. Secondary Outcome: Incidence of Closure Success
Description: Incidence of access site closure success: defined as technical success and freedom from major complications
Time Frame: Within 48 hours of the index procedure or hospital discharge, whichever occurs first
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects). Due to missing data from 2 subjects, the analysis was conducted on 112 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Transfemoral Approach: Closure of Common Femoral Artery site of subjects who have undergone interventional procedures using 8-18Fr ID sheaths.
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 112
Participants | 99

8. Secondary Outcome: Incidence of Treatment Success
Description: Incidence of Treatment Success: defined as technical success and freedom from major complications
Time Frame: 30 days post procedure
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects). Due to missing data from 3 subjects, the analysis was conducted on 111 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 111
Participants | 98

9. Secondary Outcome: Incidence of Surgical or Endovascular Intervention Post Closure
Description: Subjects requiring adjunctive surgical or endovascular intervention to achieve hemostasis of the access site (target limb only) including type of adjunctive intervention.
Time Frame: 30 days post procedure
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 110
Participants | 8

10. Secondary Outcome: Incidence of Manual Compression
Description: Incidence of subjects requiring adjunctive manual compression following use of the investigational device to achieve hemostasis of the access site (target limb only).
Time Frame: Post-procedure, following use of the investigational device until achieve hemostasis, assessed approximately up to 48 hours
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 111
Participants | 31

11. Secondary Outcome: Time-to-Ambulation:
Description: Time-to-Ambulation: defined as elapsed time from final procedural sheath removal to time when the subject stands and walks at least 20 feet without re-bleeding.
Time Frame: From the final procedural sheath removal to time when the subject stands and walks at least 20 feet without re-bleeding, assessed up to approximately 48 hours
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects). Due to missing data from 6 subjects, the analysis was conducted on 108 subjects.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 108
Hours | 15.9 (14.65)

12. Secondary Outcome: Incidence of Device Failure
Description: Incidence of subjects experiencing Device Failure.
Time Frame: 30 days post procedure
Population: Pivotal Effectiveness cohort included 114 subjects from the full analysis set, comprising all enrolled and treated without adjunctive therapy. To account for early study termination due to COVID-19 concerns, the last 18 subjects Roll-in subjects were included in the pivotal cohort (96 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 114
Participants | 0

13. Secondary Outcome: Incidence of Procedure Related Complications
Description: Number of subjects with procedure related complications as adjudicated by the CEC.
Time Frame: 30 days post procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral Approach
Number analyzed (Participants) | 88
Participants | 9

ADVERSE EVENTS:
Time Frame: From time of enrollment through study completion (up to 60 days).
Description: Evaluation of all Adverse Events (AEs) from time of investigational device use within 30 days post-procedure, and through 60 days post-procedure for subjects requiring a repeat DUS, including major and minor complications.
Arm/Group | Cross-Seal System
All-Cause Mortality (participants affected / at risk) | 1/147
Serious Adverse Events (participants affected / at risk) | 42/147
Other Adverse Events (participants affected / at risk) | 63/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cross-Seal System (N=147)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Arterial perforation (General disorders) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1) — Thoracic graft migration
Electrocardiogram PR prolongation (Investigations) | 1 (1)
Femoral artery dissection (Vascular disorders) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stent-graft endoleak (Vascular disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access site haematoma (General disorders) | 1 (1)
Vascular access site haemorrhage (General disorders) | 2 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cross-Seal System (N=147)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Anaemia postoperative (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Atheroembolism (Vascular disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Balance disorder (General disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 2 (2)
Burning sensation (General disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Carotid bruit (Investigations) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Chest discomfort (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
Ecchymosis (Vascular disorders) | 1 (1)
Ecchymosis (Blood and lymphatic system disorders) | 3 (3)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Nodule (General disorders) | 4 (4)
Oedema peripheral (Cardiac disorders) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 4 (4)
Peripheral artery thrombosis (Cardiac disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (General disorders) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Stenosis (General disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Tremor (Nervous system disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 4 (4)
Vascular access site bruising (General disorders) | 3 (3)
Vascular access site haematoma (General disorders) | 3 (3)
Vascular access site haematoma (Vascular disorders) | 2 (2)
Vascular access site haemorrhage (General disorders) | 5 (5)
Vascular access site pseudoaneurysm (General disorders) | 1 (1)
Vascular access site thrombosis (General disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03756558/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03756558/SAP_001.pdf